CLINICAL TRIAL: NCT07288385
Title: Investigating the Feasibility of Combining Virtual Reality and Bilateral Transcranial Direct Stimulation to Improve Upper Limb Recovery in Patients With Stroke
Acronym: bi-tDCS+VR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: King Saud Medical City (Other Government); King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Sarah Almhawas, PT, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB NO-25-390 KFMC; IRB NO- 25-390 (Other: IRB in King Fahad Medical City)
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Stroke; Paresis
Keywords: ischemic stroke; Hemorrhagic stroke; bi-tDCS; Hemiparesis; Neural activation; Primary motor cortex; NIBS; Non-invasive brain stimulation; Transcranial direct current stimulation; Stroke
MeSH Terms: conditions — Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Stroke; Paresis; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Intervention Model Description: Experimental: Bi-tDCS combined with VR
  20 minutes of Bi-tDCS combined with 45 minutes of VR
  Device: Transcranial Direct Current Stimulation combined with virtual reality
  20 minutes of tDCS during 45 minutes of VR games.
  Bi-tDCS will be used during the sessions. The anodal tDCS (2 mA) will be applied for 20 minutes. Continuous, direct currents. The anodal electrode will be positioned over the ipsilesional primary motor cortex (M1) of the affected hemisphere and the cathodal electrode over the contralesional hemisphere.
  Sham Comparator: tDCS+ VR
  20 minutes of sham tDCS combined with 45 minutes of VR 45 minutes of VR games with sham tDCS
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bi-tDCS+VR (Experimental): 20 minutes of tDCS during 45 minutes of VR games.
  Interventions: Device: Transcranial Direct Current Stimulation combined with virtual reality
- tDCS+ VR 20 minutes of sham tDCS combined with 45 minutes of VR (Sham Comparator)
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation combined with virtual reality — 20 minutes of tDCS during 45 minutes of VR games.
  bi-tDCS will be used during the sessions. The anodal tDCS (2 mA) will be applied for 20 minutes. Continuous, direct currents. The anodal electrode will be positioned over the ipsilesional primary motor cortex (M1) of the affected hemisphere and the cathodal electrode over the contralesional hemisphere.
  Arms: bi-tDCS+VR
Other: Sham Comparator — 45 minutes of VR games with sham tDCS. This provides the participants with the experience of the initial itchy sensation that occurs during tDCS, which is required for efficient masking.
  Arms: tDCS+ VR 20 minutes of sham tDCS combined with 45 minutes of VR

SUMMARY:
Following a stroke, the function of the distal upper limb, especially hand and finger movements, is often severely compromised, significantly restricting the ability to carry out daily activities. It is estimated that 55-75% of stroke survivors suffer from motor dysfunction, with upper limb impairments affecting up to 85% of them (Tang et al., 2024). Current rehabilitation approaches, while beneficial, often produce limited gains in hand function, particularly in patients with chronic stroke. Virtual reality (VR) training has emerged as a promising tool in neurorehabilitation, providing repetitive, task-specific, and engaging practice environments that can promote motor learning (Cameirão et al., 2012). tDCS has also shown potential to enhance motor recovery when combined with motor practice (Kang et al., 2016). To date, no studies have directly compared the effectiveness of Bi-tDCS with VR for improving upper limb function after stroke.

ELIGIBILITY:
Inclusion Criteria: 1- Adult participants (over 18 years of age) (Elsner et al., 2020).

2- Patients with a unilateral cerebral infarction or haemorrhage who are at least three months post-stroke (Muller et al., 2021).

3- Adequate mental status confirmed by an MMSE (Arabic version) should be ≥24 (Kim, 2021). ensuring the ability to comprehend and follow instructions.

4- Modified Ashworth scale score < 3 (Ögün et al., 2019). 5- Fugl-Meyer assessment (FMA) scores between 29 and 58, indicating moderate impairments (Woytowicz et al., 2017).

-

Exclusion Criteria: - Visual impairment and severe hemisensory neglect or inattention (Stahl et al., 2019; Fluet1 et al., 2015).

2- Individuals who have aphasia find it difficult to follow instructions (Fluet et al., 2015).

3- Presence of any medical condition that contraindicates the use of non-invasive brain stimulation (Stahl et al., 2019; Learmonth et al., 2021).

4- History of neurological disorders unrelated to stroke or participation in another study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-28 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test (WMFT) | at baseline and after intervention (4 weeks).
  The WMFT is a standardized assessment used to measure upper extremity motor ability through the performance of 17 tasks that include both functional and strength components. Rated using the 6-point scale ranging from 0 (no attempt) to 5 (normal movement). The total performance time and quality of movement are recorded, with lower scores indicating lower levels of functioning.
Fugl-Meyer Assessment Scale Upper Extremity (FMA-UE): | at baseline and after intervention (4 weeks).
  The FMA-UE is a comprehensive quantitative measure designed to evaluate motor function, coordination, and reflex activity of the affected upper limb following stroke. It uses a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully), with a maximum score of 66 points for the upper extremity. It is considered the gold standard for assessment of upper limb motor recovery.
Box and Block Test (BBT): | at baseline and after intervention (4 weeks).
  The BBT is a validated measure of gross manual dexterity that evaluates how many 1-inch wooden blocks a participant can transfer from one compartment to another within 60 seconds using one hand. The apparatus consists of a wooden box divided into two equal sections containing 150 small cubes. The test begins with the unaffected upper limb to allow practice and establish a baseline performance. Participants are then instructed to move as many blocks as possible, one at a time, over the partition within the time limit. The score is defined as the total number of blocks successfully transferred within 60 seconds.
Cortical Excitability Assessment: | at baseline and after intervention (4 weeks).
  Corticospinal excitability will be evaluated using transcranial magnetic stimulation (TMS) to measure motor evoked potentials (MEPs) elicited by TMS in both the affected and unaffected motor cortices (Wassermann et al., 2008). Electromyographic (EMG) activity will be monitored in real-time during TMS application, with MEPs recorded bilaterally from the first dorsal interosseous (FDI)
Functional magnetic resonance imaging (fMRI): | at baseline and after intervention (4 weeks).
  Functional magnetic resonance imaging (fMRI), a specialized form of MRI, will be utilized to assess brain activity and neural connectivity. The fMRI protocol will employ a block design paradigm, with each scanning session lasting 6 minutes and divided into six blocks. Each block will consist of 15 repetitions of 2-second contractions, separated by 30-second rest intervals (Wen et al., 2014). During the task, participants will be instructed to squeeze a rubber ball with their affected hand at an intensity corresponding to 30% of their maximum voluntary contraction force (Cheng et al., 2021; Ismail et al., 2014). Visual cues will be displayed to assist participants in achieving the target force level (Könönen et al., 2012).

SECONDARY OUTCOMES:
The Arabic version of the Stroke Specific Quality of Life Scale (SS-QOL): | at baseline and after intervention (4 weeks).
  The Stroke Specific Quality of Life Scale (SS-QOL) is a self-report questionnaire designed to assess quality of life. The 49 items on the SS-QOL measure are divided into 12 domains, which include family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity function, vision, energy, and work/productivity. Each of the 49 items is evaluated on a consistent five-point scale. Each item's responses are summed up, and the composite score that results varies from a minimum of 49 to a maximum of 245; higher scores indicate a better quality of life. The SS-QOL-49 has been translated into Arabic, and it has good validity and reliability for patients with stroke (Sallam et al., 2019).
Arabic Version of Stroke Impact Scale (SIS-16): | at baseline and after intervention (4 weeks).
  The Stroke Impact Scale (SIS) is a specific self-report measure used to assess health status in individuals after a stroke. It includes 16 items that assess different aspects of daily functioning: 7 items cover basic and instrumental activities of daily living, 8 items focus on mobility, and 1 item evaluates hand function. Each item is rated on a 5-point Likert scale, ranging from 1 (unable to complete) to 5 (no difficulty at all) (P. Duncan et al., 2003; P. W. Duncan et al., 2003). Higher scores reflect a better health-related quality of life among patients with stroke (P. W. Duncan et al., 2003). The SIS-16 is a valid and reliable tool for evaluating quality of life in patients with stroke (Chou et al., 2015).

CONTACTS AND LOCATIONS:
Locations (1):
- King Fahad Medical City مدينه الملك فهد الطبيه, 6496 Makkah Al Mukarrama Road, الرياض, الرياض 12231, Riyadh, Saudi Arabia